CLINICAL TRIAL: NCT01208090
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy, Safety & Tolerability of Two Doses of ACT-128800, an Oral S1P1 Receptor Agonist, Administered up to Twenty-eight Weeks in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: ACT-128800 in Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-058A201
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis
Keywords: psoriasis; chronic plaque psoriasis; Moderate to severe chronic plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ponesimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Investigational drug - Dose 1 (Experimental)
  Interventions: Drug: ACT-128800
- Investigational drug - Dose 2 (Experimental)
  Interventions: Drug: ACT-128800
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT-128800 — ACT-128800 (Dose 1 or Dose 2) or matching placebo administered orally once daily
  Arms: Investigational drug - Dose 1; Investigational drug - Dose 2
Drug: Placebo — ACT-128800 (Dose 1 or Dose 2) or matching placebo administered orally once daily
  Arms: Matching placebo

SUMMARY:
This study will assess the efficacy, safety and tolerability of two doses of ACT 128800 in patients with moderate-to-severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18 to 60 years (inclusive) with moderate to severe chronic plaque psoriasis who require systemic treatment.

Exclusion Criteria:

* Patients with other forms of psoriasis and patients who are currently treated for autoimmune disorders other than psoriasis.
* Systemic or topical treatments for psoriasis other than emollients. Ongoing bacterial, viral or fungal infections.

History or presence of malignancy.

* Additional inclusion and exclusion criteria apply with respect to medical conditions and concomitant treatments which could affect patients' risk from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2010-10-31 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-11-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with at least 75% improvement in PASI from baseline (PASI75) at Week 16. | Baseline to week 16

SECONDARY OUTCOMES:
Proportion of patients with "Clear" or "Almost clear" on PGA at Week 16. | Baseline to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Pharmaceuticals, Study Director — Actelion
Locations (67):
- Austria (5):
  - Clinical Investigative Site 1006, Feldkirch
  - Clinical Investigative Site 1002, Graz
  - Clinical Investigative Site 1004, Sankt Pölten
  - Clinical Investigative Site 1007, Vienna
  - Clinical Investigative Site 1001, Vienna
- Belgium (3):
  - Clinical Investigative Site 1103, Brussels
  - Clinical Investigative Site 1102, Edegem
  - Clinical Investigative Site 1101, Liège
- Bulgaria (6):
  - Clinical Investigative Site 1205, Pleven
  - Clinical Investigative Site 1204, Plovdiv
  - Clinical Investigative Site 1202, Sofia
  - Clinical Investigative Site 1201, Sofia
  - Clinical Investigative Site 1203, Sofia
  - Clinical Investigative Site 1206, Stara Zagora
- Czechia (4):
  - Clinical Investigative Site 1402, Hradec Králové
  - Clinical Investigative Site 1405, Nový Jičín
  - Clinical Investigative Site 1406, Pardubice
  - Clinical Investigative Site 1401, Prague
- Denmark (2):
  - Clinical Investigative Site 1502, Copenhagen
  - Clinical Investigative Site 1504, Roskilde
- France (7):
  - Clinical Investigative Site 1704, Bordeaux
  - Clinical Investigative Site 1701, Nice
  - Clinical Investigative Site 1707, Paris
  - Clinical Investigative Site 1710, Paris
  - Clinical Investigative Site 1705, Pierre-Bénite
  - Clinical Investigative Site 1703, Poitiers
  - Clinical Investigative Site 1702, Saint-Etienne
- Hungary (6):
  - Clinical Investigative Site 2002, Budapest
  - Clinical Investigative Site 2001, Debrecen
  - Clinical Investigative Site 2006, Miskolc
  - Clinical Investigative Site 2005, Pécs
  - Clinical Investigative Site 2003, Szeged
  - Clinical Investigative Site 2004, Veszprém
- Italy (8):
  - Clinical Investigative Site 2315, Ancona
  - Clinical Investigative Site 2303, Bergamo
  - Clinical Investigative Site 2307, Bologna
  - Clinical Investigative Site 2317, Genova
  - Clinical Investigative Site 2309, L’Aquila
  - Clinical Investigative Site 2310, Pisa
  - Clinical Investigative Site 2304, Roma
  - Clinical Investigative Site 2316, Rome
- Clinical Investigative Site 3801, Vilnius, Lithuania
- Romania (8):
  - Clinical Investigative Site 2608, Bucharest
  - Clinical Investigative Site 2601, Bucharest
  - Clinical Investigative Site 2604, Cluj-Napoca
  - Clinical Investigative Site 2603, Iași
  - Clinical Investigative Site 2606, Oradea
  - Clinical Investigative Site 2607, Sibiu
  - Clinical Investigative Site 2605, Târgu Mureş
  - Clinical Investigative Site 2602, Timișoara
- Clinical Investigative Site 3410, Krasnodar, Russia
- Slovakia (4):
  - Clinical Investigative Site 2704, Banská Bystrica
  - Clinical Investigative Site 2705, Kosice-Saca
  - Clinical Investigative Site 2701, Košice
  - Clinical Investigative Site 2708, Trnava
- Spain (4):
  - Clinical Investigative Site 2901, Barcelona
  - Clinical Investigative Site 2907, Las Palmas de Gran Canaria
  - Clinical Investigative Site 2902, Madrid
  - Clinical Investigative Site 2904, Madrid
- Sweden (2):
  - Clinical Investigative Site 3001, Stockholm
  - Clinical Investigative Site 3006, Umeå
- Switzerland (2):
  - Clinical Investigative Site 3101, Lausanne
  - Clinical Investigative Site 3103, Zurich
- Ukraine (2):
  - Clinical Investigative Site 3512, Poltava
  - Clinical Investigative Site 3514, Zaporizhia
- United Kingdom (2):
  - Clinical Investigative Site 3306, Dundee
  - Clinical Investigative Site 3304, London

REFERENCES:
- [Derived] Vaclavkova A, Chimenti S, Arenberger P, Hollo P, Sator PG, Burcklen M, Stefani M, D'Ambrosio D. Oral ponesimod in patients with chronic plaque psoriasis: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet. 2014 Dec 6;384(9959):2036-45. doi: 10.1016/S0140-6736(14)60803-5. Epub 2014 Aug 10. PMID 25127208